CLINICAL TRIAL: NCT03628937
Title: The Effect of Decaffeinated Green Tea Polyphenol Intake on the Risk of Precocious Puberty Among Obese Girls
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XH-18-009
Record Dates: First submitted 2018-07-10; First posted 2018-08-14 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2019-12

CONDITIONS: Pediatric Obesity; Puberty, Precocious
Keywords: Green tea polyphenols; Children obesity; Precocious puberty; Prevention
MeSH Terms: conditions — Pediatric Obesity; Puberty, Precocious

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Interventions: Decaffeinated green tea polyphenol capsule (400 mg, EGCG accounted for 50%) will be given to participants in intervention group, and they need take it once a day after breakfast for 12 weeks.
  Decaffeinated green tea polyphenol: 400mg/capsule, 1 capsule/d, qd, 12 weeks
  Interventions: Dietary Supplement: Decaffeinated Green Tea Polyphenol
- Control group (Placebo Comparator): The placebo control group will be given placebo capsules, and participants need take it once a day after breakfast for 12 weeks.
  Interventions: Other: Placebo control

INTERVENTIONS:
Dietary Supplement: Decaffeinated Green Tea Polyphenol — Intervention group will be given decaffeinated green tea polyphenol capsules (400 mg, EGCG accounted for 50%). Participants need take it once a day after breakfast for 12 weeks.
  Arms: Intervention group
Other: Placebo control — The starch capsule was used as a placebo control, which has the same dosage, appearance and smell compared to decaffeinated green tea polyphenol capsule. The use frequency and duration are consistent with intervention group.
  Arms: Control group

SUMMARY:
In this study, 6-10 years old obese girls will be recruited to test the preventive effect of decaffeinated green tea polyphenols on the risk of precocious puberty by the random, placebo-control and single blind design. The intervention group will be given decaffeinated green tea polyphenols capsule (400mg/d) and the control group will be given placebo. The oral treatment will be lasted for 12 weeks.Then all the subjects will be followed up every 3 months until three months after menstruation. At the baseline and after the 12 week intervention, the clinical manifestations of secondary sexual characters, the serum levels of sex hormones will be determined as the outcome variables. After controlling confounding factors, the preventive effect of the green tea polyphenols on precocious puberty or early puberty among obese girls will be analyzed.

DETAILED DESCRIPTION:
Simple obese girls are prone to premature or early puberty. The topic proposed based on previous studies, recruiting of 80 simple overweight or obesity girls, aged 6 to 10 years old. After the informed consent, they will be randomly divided into intervention group and control group, intervention group will be given tea polyphenol capsule (400 mg, epigallocatechin gallate (EGCG) accounted for 50%), the control group given placebo capsule. Participants need take it once a day after breakfast. All of them will receive similar health advice on proper diet and exercise. The intervention will last 12 weeks, followed by telephone every 3 months until 3 months after menarche. The researchers will measure children obesity index (using artificial detection), youth development index (secondary sex characteristic clinical manifestations, serum sex hormone, B ultrasonic examination uterus ovarian and breast volume, etc.) in three stages: at the baseline, after 12 weeks intervention and the end of three months after menstruation. The liver and kidney function, blood and urine routine and serum trace elements will be detected before and after the three-month intervention. Through the above detection of the indicators related to obesity and sexual precocious puberty, it is explored whether the decaffeinated tea polyphenol has preventive effects on precocious puberty.

ELIGIBILITY:
Inclusion Criteria:

1. 6-10 years old;
2. BMI reached or exceeded the overweight or obesity threshold of school-aged girls in China (6 years old, BMI>=16.3; 7 years old, BMI>=17.2; 8 years old, BMI>=18.1;9 years old, BMI>=19.0; Age of 10, BMI>=20.0);
3. having not received sex hormone drugs, gonadotropin-releasing hormone (GnRH) drugs and Chinese medicine for the prevention and treatment of precocious puberty in the past;
4. the guardian's informed consent;

Exclusion Criteria:

1. secondary obesity (such as hormone therapy);
2. weight loss treatment is currently under way;
3. menarche or central precocious puberty has been clearly diagnosed;
4. patients with serious heart, liver, kidney, hematopoietic system diseases and endocrine genetic metabolic diseases;
5. iron therapy is under way;
6. patients with acute and chronic inflammation;
7. other conditions that the researchers believe may influence the observation results.

Ages: 6 Years to 10 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of Precoicous Puberty in the intervention groups and the placebo group. | about two years
  Female precocious puberty is defined as the development of secondary sexual characteristics before the age of 8 or menarche before the age of 10. In our study, after intervention, for girls under 8 years of age, we recorded their rate of secondary sexual characteristics at 8 years of age; and for girls under 10 years of age, we recorded their rate of menarche at 10 years of age. The difference in the incidence of precocious puberty between the two groups is the primary outcome.

SECONDARY OUTCOMES:
The average age of onset of menarche in two groups | an average of 4 years
  Record the age of the onset of menarche of each girl and comparing the average age between two groups, to explore whether green tea polyphenols could delay the early pubertal development.
The change in BMI at week 12 intervention from the baseline | 12 weeks
  Obesity is an important contributing factor to the early onset of puberty for girls. Green tea polyphenols may prevent precocious puberty by controlling body weight and reducing serum leptin level.
The change of breast tissue volume at week 12 intervention from the baseline | 12 weeks
  These indicator is important indicators related to sexual development.
The change of uterus volume at week 12 intervention from the baseline | 12 weeks
  These indicator is important indicators related to sexual development.
The change of the number of follicles with diameter of > 4mm follicles in ovary at week 12 intervention from the baseline | 12 weeks
  These indicator is important indicators related to sexual development.
The change of serum sex hormone levels at week 12 intervention from the baseline | 12 weeks
  These indicators are important indicators related to sexual development.
The status of liver and kidney function at the baseline and after 12 weeks intervention | 12 weeks
  To identify the safety of green tea polyphenol intake for obese girls

CONTACTS AND LOCATIONS:
Overall Officials: Xiuhua Shen, Professor, Study Chair — Xinhua Hospital Afflicated to Shanghai Jiaotong University of Medicine
Locations (1):
- Department of Clinical Nutrition, Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xie L, Tang Q, Yao D, Gu Q, Zheng H, Wang X, Yu Z, Shen X. Effect of Decaffeinated Green Tea Polyphenols on Body Fat and Precocious Puberty in Obese Girls: A Randomized Controlled Trial. Front Endocrinol (Lausanne). 2021 Oct 12;12:736724. doi: 10.3389/fendo.2021.736724. eCollection 2021. PMID 34712203